CLINICAL TRIAL: NCT02464670
Title: Phase 1, Open-Label Study to Evaluate the Safety, Tolerability, and Immunogenicity of INO-4212 and Its Components, INO-4201 and INO-4202, Given With or Without INO-9012, Administered IM or ID Followed by Electroporation in Healthy Volunteers
Brief Title: Open-Label Study of INO-4212 With or Without INO-9012, Administered IM or ID Followed by Electroporation in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Collaborators: GeneOne Life Science, Inc. (Industry); Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: EBOV-001
Record Dates: First submitted 2015-05-28; First posted 2015-06-08 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Ebola Vaccine
Keywords: Ebola; Vaccine
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — rocakinogene sifuplasmid

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: In Part II only (Groups 3A and 3B), the current strength of the device will be masked from the study team administering the procedure and participant. All IP assignments will be open label and unmasked.
Oversight: Data Monitoring Committee: No

ARMS (13):
- Group 1 (Experimental): INO-4201 IM + EP, 2 mg, 3 doses
  Interventions: Biological: INO-4201
- Group 2 (Experimental): INO-4202 IM + EP, 2 mg, 3 doses
  Interventions: Biological: INO-4202
- Group 3 (Experimental): INO-4201 ID + EP 0.2A, 2 mg, 3 doses
  Interventions: Biological: INO-4201
- Group 4 (Experimental): INO-4212 IM + EP, 4 mg, 3 doses
  Interventions: Biological: INO-4212
- Group 5 (Experimental): INO-4212 + INO-9012 IM + EP, 4+1 mg, 3 doses
  Interventions: Biological: INO-4212 + INO-9012
- Group 6 (Experimental): INO-4201 ID + EP 0.2A, 1 mg, 3 doses
  Interventions: Biological: INO-4201
- Group 7 (Experimental): INO-4201 ID + EP 0.2A, 2 mg, 2 doses
  Interventions: Biological: INO-4201
- Group 8 (Experimental): INO-4201 ID + EP 0.2A, 1 mg, 2 doses
  Interventions: Biological: INO-4201
- Group 9 (Experimental): INO-4201 + INO-9012 ID + EP 0.2A, 1.6 + 0.4 mg, 3 doses
  Interventions: Biological: INO-4201 + INO-9012
- Group 10 (Experimental): INO-4201 + INO-9012 ID + EP 0.2A, 1.6 + 0.4 mg, 2 doses
  Interventions: Biological: INO-4201 + INO-9012
- Group 11 (Experimental): INO-4201 + INO-9012 ID + EP 0.2A, 0.8 + 0.2 mg, 3 doses
  Interventions: Biological: INO-4201 + INO-9012
- Part II: Group 3A (Experimental): INO-4201 ID + EP 0.2A, 2 mg, 3 doses
  Interventions: Biological: INO-4201
- Part II: Group 3B (Experimental): INO-4201 ID + EP 0.1A, 2 mg, 3 doses
  Interventions: Biological: INO-4201

INTERVENTIONS:
Biological: INO-4201 — INO-4201 delivered IM followed by Electroporation
  Arms: Group 1
Biological: INO-4202 — INO-4202 delivered IM followed by Electroporation
  Arms: Group 2
Biological: INO-4201 — INO-4201 delivered ID followed by Electroporation
  Arms: Group 3; Group 6; Group 7; Group 8; Part II: Group 3A; Part II: Group 3B
Biological: INO-4212 — INO-4212 delivered IM followed by Electroporation
  Arms: Group 4
Biological: INO-4212 + INO-9012 — INO-4212 + INO-9012 delivered IM followed by Electroporation
  Arms: Group 5
Biological: INO-4201 + INO-9012 — INO-4201 + INO-9012 delivered ID followed by Electroporation
  Arms: Group 10; Group 11; Group 9

SUMMARY:
This study evaluates whether INO-4212 and its components INO-4201 and INO-4202 administered intramuscularly (IM) or intradermally (ID) followed by electroporation (EP) will be well tolerated and immunogenic.

DETAILED DESCRIPTION:
This study will test the safety, tolerability, and immunogenicity of the DNA vaccine, INO-4212 and its components INO-4201 and INO-4202 in healthy volunteers. INO-4201 contains the DNA sequence that codes for past Ebola Zaire virus outbreak strains, and INO-4202 contains the DNA sequence that codes for the current Ebola virus outbreak strain. When given together, the DNA vaccine is called INO-4212 and contains the DNA sequence of both the previous and the current outbreak strain. Another ingredient called INO-9012 which contains the DNA sequence for interleukin-12, will be given in a subset of subjects to help boost the body's immune response when given with the vaccine.

Following administration of vaccine, a specialized medical device, CELLECTRA®, will deliver brief electrical pulses in a process known as electroporation (EP), to help move more DNA into cells more efficiently. The study will evaluate whether INO-4212 and its components may be able to generate protective immunity against Ebola Zaire, evaluate the relative ability of IM versus ID administration to elicit immune responses and evaluate whether vaccine administered with INO-9012 can generate greater immune responses.

The Ebola vaccine under study will be tested in approximately 240 healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years;
* Able to provide consent to participate and having signed an Informed Consent Form (ICF);
* Able and willing to comply with all study procedures;
* Women of child-bearing potential who are in a relationship that could result in pregnancy agree to either remain sexually abstinent, use medically effective contraception (oral contraception, barrier methods, spermicide, etc.) or have a partner who is sterile from enrollment to 3 months following the last injection; OR, sexually active men who are considered sexually fertile must agree to use either a barrier method of contraception during the study, and agree to continue the use for at least 3 months following the last injection, or have a partner who is permanently sterile or unable to become pregnant;
* Normal screening ECG or screening ECG with no clinically significant findings;
* Screening laboratory (Complete blood count (CBC), serum electrolytes, blood urea nitrogen (BUN), creatinine (Cr), glucose, ALT, CPK, urinalysis) grade 0-1 within 30 days prior to administration of study treatment;
* No history of clinically significant immunosuppressive or autoimmune disease.

Exclusion Criteria:

* Administration of an investigational compound either currently or within 30 days of first dose;
* Previous receipt of an investigational product in an interventional trial for the treatment or prevention of Ebola (exceptions: verified receipt of placebo only or participation in an observational study);
* History of or positive serologic test for HIV, hepatitis B surface antigen (HBsAg); or any potentially communicable infectious disease as determined by the Principal Investigator or Medical Monitor;
* Positive serologic test for hepatitis C (exception: successful treatment with confirmation of sustained virologic response);
* Baseline creatinine greater than 1.5 (CKD Stage II or greater);
* Chronic liver disease or cirrhosis;
* Immunosuppressive illness including hematologic malignancy, history of solid organ or bone marrow transplantation;
* Any pre-excitation syndromes, e.g., Wolff-Parkinson-White syndrome;
* Prior major surgery or radiation therapy within 4 weeks of randomization;
* Pregnant, breast feeding, or considering becoming pregnant;
* Less than two acceptable sites exist for intramuscular or intradermal injection and EP between use of the deltoid and lateral quadriceps muscles. A site for injection/EP is not acceptable if there are tattoos, keloids or hypertrophic scars within 2 cm of the injection/EP site.
* Subject has significant acute or chronic medical illness if deemed by the practitioner that electroporation treatment could negatively impact the illness
* Subject has unstable or life-threatening cardiac disease (e.g. unstable angina, class 3 or higher congestive heart failure)
* Subject has an acute or chronic bleeding or clotting disorder that would contraindicate IM injections or use of blood thinners (e.g. anticoagulants or antiplatelet drugs) within 2 weeks;
* Subject has a cardioverter-defibrillator or pacemaker (to prevent a life-threatening arrhythmia) that is located ipsilateral to the intended deltoid injection site (unless deemed acceptable by a Cardiologist);
* Subject has metal implant or implantable medical device within the electroporation area;
* Administration of any vaccine within 4 weeks of first dose;
* Administration of any blood product within 3 months of first dose;
* Current or anticipated concomitant immunosuppressive therapy (excluding inhaled, topical skin and/or eye drop-containing corticosteroids, or low-dose methotrexate). Systemic corticosteroids must be discontinued at least 4 weeks prior to first dose;
* Current or anticipated treatment with TNF-α inhibitors such as infliximab, adalimumab, etanercept;
* Active military service personnel;
* Prisoner or subjects who are compulsorily detained (involuntary incarceration) for treatment of either a physical or psychiatric illness;
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements or assessment of immunologic endpoints; or
* Any illness or condition that in the opinion of the investigator may affect the safety of the subject or the evaluation of any study endpoint.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2015-05; Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Safety Assessment (Composite of multiple measures: adverse events, pain (VAS), lab abnormalities, changes in vital signs) | Screening through up to 60 weeks following the first dose
  Composite of multiple measures consist of:
  * Frequency and severity of all adverse events
  * Local pain immediately and at 5 and 10 minutes after Study Treatment/EP using a visual analog scale from 0 to 10, with 0 representing "No Pain" and 10 representing "Worst Pain"
  * Frequency and severity of local and systemic events for at least 7 days after Study Treatment/EP
  * Frequency and severity of laboratory abnormalities
  * Changes in vital signs (blood pressure, heart rate, respiratory rate, temperature)

SECONDARY OUTCOMES:
Immunology Assessment | Screening and at select points up to 60 weeks following the first dose
  Composite outcome measure consisting of multiple measures, including:
  * Breadth and magnitude of antigen specific ELISA
  * Breadth and magnitude of neutralizing antibodies
  * Breadth and magnitude of antigen specific cellular immune responses as determined by
    * Interferon-gamma (IFN-γ) ELISpot
    * Intracellular Cytokine Staining (CTL phenotype, Lytic granule loading, Granzyme B killing of target cells)

OTHER OUTCOMES:
Exploratory Assessment | Screening and at select points up to 60 weeks following the first dose
  Composite outcome measure consisting of multiple measures, including:
  * Differences in immune response between ID delivery of INO-4201 followed by EP compared to IM delivery of INO-4201 followed by EP
  * Differences in immune response between IM delivery of INO-4212 in combination with INO-9012 followed by EP compared to IM delivery of INO-4212 alone followed by EP
  * Differences in immune response between ID delivery of INO-4201 in combination with INO-9012 followed by EP compared to ID delivery of INO-4201 alone followed by EP
  * Differences in immune response between 2 doses or 3 doses of INO-4201 alone or in combination with INO-9012 administered ID followed by EP
  * Differences in immune response between either 1 mg or 2mg total of INO-4201 alone or in combination with INO-9012 administered ID followed by EP
  * Differences in immune response between ID delivery of INO-4201 followed by EP with either 0.2 A or 0.1 A
  * Perception of injection among subjects enrolled in Part II

CONTACTS AND LOCATIONS:
Overall Officials: Scott White, MD, Study Director — Inovio Pharmaceuticals
Locations (3):
- United States (3):
  - QPS MRA, Miami, Florida
  - The Center for Pharmaceutical Research, Kansas City, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Tebas P, Kraynyak KA, Patel A, Maslow JN, Morrow MP, Sylvester AJ, Knoblock D, Gillespie E, Amante D, Racine T, McMullan T, Jeong M, Roberts CC, Park YK, Boyer J, Broderick KE, Kobinger GP, Bagarazzi M, Weiner DB, Sardesai NY, White SM. Intradermal SynCon(R) Ebola GP DNA Vaccine Is Temperature Stable and Safely Demonstrates Cellular and Humoral Immunogenicity Advantages in Healthy Volunteers. J Infect Dis. 2019 Jul 2;220(3):400-410. doi: 10.1093/infdis/jiz132. PMID 30891607